CLINICAL TRIAL: NCT02440763
Title: The EUROSCA Natural History Study
Acronym: EUROSCA-NHS
Status: Recruiting | Type: Observational
Sponsor: Ataxia Study Group (Other)
Responsible Party: Sponsor
Other Study IDs: 010/05
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Spinocerebellar Ataxia
Keywords: Natural History
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA is obtained for genetic testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinocerebellar ataxia type 1,2,3 and 6: Spinocerebellar ataxias (SCA) are autosomal dominantly inherited progressive ataxia disorders. An epidemiological study performed in the Netherlands found a prevalence of 3.0 : 100,000 (van de Warrenburg et al. 2002). The SCA´s are genetically and clinically heterogeneous disorders with SCA1, SCA2, SCA3 and SCA6 being the most frequent genotypes worldwide. While SCA1, SCA2 and SCA3 have a complex phenotype, SCA6 patients usually present with pure cerebellar ataxia (Schols et al. 2004). Although precise knowledge of the rate of disease progression is a prerequisite for the biometrical design of future therapeutical trials, prospective studies of the natural history of SCA´s have not been performed. Similarly, the occurrence and evolution of accompanying non-ataxia symptoms have not been studied prospectively.

SUMMARY:
The key goals of EUROSCA-NHS is to determine and compare the rate of disease progression in SCA1, SCA2, SCA3 and SCA6 including determination of the order and occurrence of non-ataxia symptoms, assessment of activities of daily living (ADL) and quality of life (QoL), and identification of predictors of disease progression and survival.

DETAILED DESCRIPTION:
The key goal of EUROSCA-NHS is to determine and compare the rate of disease progression in SCA1, SCA2, SCA3 and SCA6. To this end, a newly developed and validated ataxia scale (Scale for the Assessment and Rating of Ataxia, SARA) will be used. EUROSCA-NHS has a number of secondary aims including determination of the order and occurrence of non-ataxia symptoms, assessment of activities of daily living (ADL) and quality of life (QoL), and identification of predictors of disease progression and survival. Substudies will deal with the development of brain atrophy, as assessed by magnetic resonance imaging (MRI), progression of peripheral neuropathy, as assessed by nerve conduction studies, and specific clinical aspects of SCA.

ELIGIBILITY:
Inclusion criteria:

* Progressive, otherwise unexplained ataxia
* Positive genetic testing for SCA1, SCA2, SCA3, and SCA6
* Written informed consent by the patient or his legal agent

Exclusion criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spinocerebellar ataxia type 1,2,3 and 6.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2005-07; Primary Completion 2050-07 (Estimated); Study Completion 2050-07 (Estimated)

PRIMARY OUTCOMES:
Scale for the assessment and rating of ataxia (SARA) | Patients are first seen at a baseline visit, followed by annual visits for 3 years scheduled ± 3 months around the specified time point. After the initial 3 year observation period, visits are done at irregular intervals each time they went to hospital.
  Progression of ataxia is measured using a newly developed and validated ataxia scale, SARA. SARA was evaluated in two large validation trials performed by the EUROSCA clinical group and was found to be easy to use, reliable, and valid.

SECONDARY OUTCOMES:
Disease stages | Patients are first seen at a baseline visit, followed by annual visits for 3 years scheduled ± 3 months around the specified time point. After the initial 3 year observation period, visits are done at irregular intervals each time they went to hospital.
  Disease stages are measured using the 5 point scale ranging from 0 to 4 proposed by Klockgether et al., 1998.
Inventory of non-ataxia signs (INAS) | Patients are first seen at a baseline visit, followed by annual visits for 3 years scheduled ± 3 months around the specified time point. After the initial 3 year observation period, visits are done at irregular intervals each time they went to hospital.
  The occurrence of accompanying non-ataxia symptoms is recorded using INAS. In the SARA validation trials, INAS was applied to a large number of SCA patients. Statistical evaluation showed good reliability.
UHDRS part IV | Patients are first seen at a baseline visit, followed by annual visits for 3 years scheduled ± 3 months around the specified time point. After the initial 3 year observation period, visits are done at irregular intervals each time they went to hospital.
  Functional disability in ADL is assessed using the Functional assessment part of the Unified Huntington's Disease Rating Scale (UHDRS) (Huntington Study Group, 1996). This 25-item assessment has been used in SCA patients throughout the SARA validation study with good practicality.
EQ-5D | Patients are first seen at a baseline visit, followed by annual visits for 3 years scheduled ± 3 months around the specified time point. After the initial 3 year observation period, visits are done at irregular intervals each time they went to hospital.
  Health related Quality of life is assessed using EQ-5D, a generic instrument that has been developed and validated by the EuroQuol Group (1990) and is available in validated translations for use as a questionnaire.
PHQ-9 | Patients are first seen at a baseline visit, followed by annual visits for 3 years scheduled ± 3 months around the specified time point. After the initial 3 year observation period, visits are done at irregular intervals each time they went to hospital.
  Assessment of depressive symptoms is done using a validated 9-item short form of the Patient Health Questionnaire (PHQ), a questionnaire that has been developed to screen for psychiatric co-morbidity in unselected populations (Spitzer et al. 1999).

CONTACTS AND LOCATIONS:
Locations (16):
- Department of Neurology, Medical University, Innsbruck, Innsbruck, Austria
- Université Libre de Bruxelles (ULB), Neurology Service - ULB Hôpital Erasme, ULB Laboratory of Experimental Neurology, Brussels, Belgium
- Hôpital de la Pitié-Salpêtrière, Département de Génétique, Paris, France
- Germany (5):
  - Department of Neurology, St. Josef Hospital, University Hospital of Bochum, Bochum
  - Department of Neurology, University of Bonn, Bonn
  - Department of Neurology, University Clinic Essen, University of Duisburg-Essen, Essen
  - Department of Neurology, University of Frankfurt, Frankfurt
  - Department of Neurodegeneration and Hertie-Institute for Clinical Brain Research, University of Tübingen, Tübingen
- Hungary (2):
  - Department of Medical Genetics, University of Pecs, Pécs
  - Department of Neurology, Zala County Hospital, Zalaegerszeg
- Italy (2):
  - Fondazione-IRCCS Istituto Neurologico Carlo Besta, Milan
  - Department of Neuroscience, Federico II University Naples, Naples
- Radboud University Medical Center, Department of Neurology, Donders Institute for Brain, Cognition, and Behaviour, Nijmegen, Netherlands
- Institute of Psychiatry and Neurology, Warsaw, Poland
- University Hospital Marqués de Valdecilla (IDIVAL), University of Cantabria, Santander, Spain
- Institute of Neurology, London, United Kingdom

REFERENCES:
- [Derived] Diallo A, Jacobi H, Cook A, Labrum R, Durr A, Brice A, Charles P, Marelli C, Mariotti C, Nanetti L, Panzeri M, Rakowicz M, Sobanska A, Sulek A, Schmitz-Hubsch T, Schols L, Hengel H, Melegh B, Filla A, Antenora A, Infante J, Berciano J, van de Warrenburg BP, Timmann D, Boesch S, Pandolfo M, Schulz JB, Bauer P, Giunti P, Kang JS, Klockgether T, Tezenas du Montcel S. Survival in patients with spinocerebellar ataxia types 1, 2, 3, and 6 (EUROSCA): a longitudinal cohort study. Lancet Neurol. 2018 Apr;17(4):327-334. doi: 10.1016/S1474-4422(18)30042-5. Epub 2018 Mar 13. PMID 29553382
- [Derived] Jacobi H, du Montcel ST, Bauer P, Giunti P, Cook A, Labrum R, Parkinson MH, Durr A, Brice A, Charles P, Marelli C, Mariotti C, Nanetti L, Panzeri M, Rakowicz M, Sulek A, Sobanska A, Schmitz-Hubsch T, Schols L, Hengel H, Baliko L, Melegh B, Filla A, Antenora A, Infante J, Berciano J, van de Warrenburg BP, Timmann D, Szymanski S, Boesch S, Kang JS, Pandolfo M, Schulz JB, Molho S, Diallo A, Klockgether T. Long-term disease progression in spinocerebellar ataxia types 1, 2, 3, and 6: a longitudinal cohort study. Lancet Neurol. 2015 Nov;14(11):1101-8. doi: 10.1016/S1474-4422(15)00202-1. Epub 2015 Sep 13. PMID 26377379